CLINICAL TRIAL: NCT06506279
Title: Motor Recovery Through Plasticity-Inducing Cortical Stimulation
Acronym: MRPICS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Jeffrey Ojemann, Professor, Neurological Surgery, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00019577; UH3NS121565 (NIH)
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Motor Recovery through Plasticity-Inducing Cortical Stimulation (Experimental): Single arm study of post-ischemic stroke patients with an upper extremity deficit.
  Interventions: Device: CorTec Brain Interchange (BIC) System

INTERVENTIONS:
Device: CorTec Brain Interchange (BIC) System — Surgical implantation of the BIC System. This study's main objective is to implement and evaluate neuroplasticity-inducing stimulation. The stimulation methods for inducing neuroplasticity have been selected based on prior preclinical and intraoperative work that has shown promise in providing rehabilitative benefits for stroke patients.

SUMMARY:
Using the CorTec Brain Interchange (BIC) System, we will examine the effect of a plasticity-inducing therapy regime on the rehabilitation of upper limb impairment post-stroke. This study's main objective is to implement and evaluate neuroplasticity-inducing stimulation. The stimulation methods for inducing neuroplasticity have been selected based on prior preclinical and intraoperative work that has shown promise in providing rehabilitative benefits for stroke patients. We will be structuring this study as an open prospective feasibility study.

DETAILED DESCRIPTION:
Stroke is one of the top three causes of human disability. In middle- and high-income countries around the world, stroke is the leading neurological cause of lost disability-adjusted life years. Motor deficits are among the most common results of stroke and contribute substantially to post-stroke disability. An estimated 6,600,000 American adults have had a symptomatic stroke, with a prevalence that increases with age. Each year, 795,000 people experience a stroke, of which 610,000 are first-ever symptomatic strokes. The mean survival after stroke is 6-7 years, with approximately 85% of patients living past the first year of stroke. With the decline in stroke mortality accompanying advances in acute stroke care and aging of the population, the disease burden is projected to increase. Thus, most patients survive their stroke and live with enduring disability for years to come.

Between 55% and 75% of patients have enduring motor deficits after stroke, which are associated with reduced quality of life, and 65% of patients at 6 months are unable to incorporate the affected hand effectively into daily activities. Subjective well-being is decreased one year after stroke, and some research attributes this decrease directly to arm motor impairments. In the long term after a stroke, at least half of patients have to rely on human assistance for basic activities of daily living (ADLs) such as feeding, self-care, and mobility. Upper extremity function is a key part of this disability after stroke. Needs assessments from patients include expectations of recovery, occupation-specific needs that may require strength vs fine motor skills, and activities of daily living, all of which will reduce overall disability measures. Upper extremity function (as measured by the Wolf Motor Function Test [WMFT]) has been shown as a predictor of quality-of-life scores.

Current therapies for a new stroke reduce disability in only a subset of patients. The only drug approved to treat acute ischemic stroke remains tissue plasminogen activator (tPA). Only a minor fraction of patients receive this medicine in large part due to the narrow time window for safe drug administration. The fraction of patients who receive endovascular therapy is even smaller. Moreover, of those so treated, half or more have significant long-term disability.

Physical therapy remains the mainstay of treatment, and advances in remote teletherapy and other home or gaming options may further increase its utilization. Non-invasive exoskeleton use has also been approved for upper extremity therapy. These existing approaches to rehabilitation have been used for decades and are widely recognized to provide important benefits. Nevertheless, the efficacy of these rehabilitation approaches is equally widely recognized to be limited such that some patients do not respond to rehabilitation, and some only show partial recovery. These important limitations in the efficacy of existing rehabilitation approaches are likely due to the very nature of physical rehabilitation: they engage peripheral nerves and muscles and likely only have indirect effects on damaged physiology in the brain. It is equally expected that direct and targeted manipulation of brain physiology has the potential to rehabilitate people with chronic stroke more effectively. Thus, there has been a growing interest in using electric or magnetic stimulation of the cortex or cortical pathways to promote brain recovery and to enhance structural and functional brain plasticity.

The study proposes to investigate the effectiveness of promoting interactions between affected and intact cortical regions by inducing neural plasticity through specific protocols. By inducing plasticity through the use of closed-loop stimulation delivered simultaneously with conventional activity-based therapy, the study results are expected to enhance recovery beyond what is achievable with therapy alone.

ELIGIBILITY:
Inclusion Criteria:

22-75 years of age

* History of ischemic stroke
* Minimum 6 months post-ischemic cortical stroke
* Levels of hemiparesis that warrant surgical intervention (upper limb impairment)
* Able to participate in a meaningful way in rehabilitation (defined by upper extremity Fugl-Myer (UEFM) score of 25-45
* Disability measured between 3 and 4 on the modified Rankin Scale
* Minimum of 30% preservation of the corticospinal pathways in MRI imaging
* Observable motor output of the upper limb in response to TMS delivered to the motor cortex
* Available for the duration of the study, 54 weeks for multiple visits (38 weeks implanted and 16 weeks post-explant follow-up).
* All inclusion and exclusion criteria will be assessed within 90 days before the device implantation procedure (though the PI may determine to override the 90-day limit for MRI imaging results review).

Exclusion Criteria:

* Unable to discontinue anti-platelet medication for 7 days pre- and 3 days post-op
* On therapeutic anticoagulation
* A history of unprovoked deep vein thrombosis or any pulmonary embolus
* The presence of a bleeding disorder which significantly increases the chances that the patient will have a hemorrhagic complication in relation to study procedures.
* Other medical history indicating increased risk of thrombosis per investigator discretion
* Any history of seizures
* Pregnancy
* Geriatric Depression Score greater than 10
* Montreal Cognitive Assessment below 22 unless attributable to aphasia and approved by PI
* Columbia Suicide Scale ideation score above 1
* Aphasia or cognitive deficits substantial enough to prevent:

  * communication of pain and discomfort due to study procedures
  * understanding of motor testing or rehabilitation tasks
* Severe Neglect as measured by NIH Stroke Scale Question 11 score of 2, which represents a "Profound hemi-inattention or extinction to more than one modality; does not recognize own hand or orients to only one side of space."
* Cardiac morbidity that in the judgment of the investigators would represent an increased safety risk
* History of spontaneous hemorrhagic stroke
* Major, active neurological, psychiatric, or medical comorbidity that would likely interfere with study procedures
* Any active infection requiring antimicrobial therapy
* Inability to participate with proposed rehabilitation strategies
* Presence of any other implanted devices (cochlear implants, pacemakers, etc.).
* During this study no occupational, physical, or speech therapy is permitted apart from that provided by the study protocol. Patients who require therapy beyond what is delivered in this study will not be enrolled
* All inclusion and exclusion criteria will be assessed within 90 days before the device implantation procedure (though the PI may determine to override the 90-day limit for MRI imaging results review).

If a patient has glenohumeral subluxation, adhesive capsulitis, or contractures of the upper extremities, they must undergo additional screening for pain with range-of-motion and be approved by the enrolling clinician.

If a patient requires any medication not already explicitly excluded as part of defined safety criteria, the clinical staff affiliated with this study will determine if the patient should be excluded at their own discretion to ensure the integrity of this study.

-

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2028-06-15 (Estimated); Study Completion 2030-06-15 (Estimated)

PRIMARY OUTCOMES:
Measuring upper limb impairment in stroke rehabilitation | Two years
  The primary outcome measure in the study focus on measuring upper limb impairment to ensure that the use of the CorTec Brain Interchange system is not detrimental for use in studying stimulation paradigms to improve stroke rehabilitation. Limb impairment will be assessed for all patients weekly during the rehabilitation period and at all monthly post-rehab monitoring visits using the primary behavioral measures of the study, UEFM (Upper Extremity Fuegl-Myer) arm motor score and the WMFT (Wolf Motor Function Test), which will track individual trends of motor improvement and motor function, respectively. In four subjects the degree of potentially confounding variables (such as injury and/or patient variability) will likely inhibit extrapolation of therapeutic outcomes to the stroke population at large.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Ojemann, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States